CLINICAL TRIAL: NCT03816189
Title: Role of Blood and Tissue Eosinophils in the Fibrogenesis of Systemic Sclerosis
Brief Title: Role of Eosinophil in Fibrogenesis of Systemic Sclerosis
Acronym: EOFIB-SSC
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 2017_10; 2017-A02587-46 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-12-18; First posted 2019-01-25 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Systemic Sclerosis; Systemic Scleroderma
Keywords: Eosinophil; Fibrosis; Systemic Scleroderma
MeSH Terms: conditions — Scleroderma, Systemic; Fibrosis | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, Eosinophils, tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Diffuse SSc: Recruitment of 20 patients with diffuse SSc
  Interventions: Diagnostic Test: Blood test; Diagnostic Test: Skin biopsies
- Limited SSc: Recruitment of 20 patients with limited SSc
  Interventions: Diagnostic Test: Blood test; Diagnostic Test: Skin biopsies
- Healthy subjects: Recruitment of 20 healthy subjects (control)
  Interventions: Diagnostic Test: Blood test

INTERVENTIONS:
Diagnostic Test: Blood test — Patients in each group will have a blood sample (9x7 mL) for eosinophils isolation, study of activation markers on whole blood and serum biomarkers testing
Diagnostic Test: Skin biopsies — In patients who will accept, skin biopsies will be performed in damaged and apparently normal skin, excluding fingers, hands, feet and face (biopsies are facultative)
  Groups: Diffuse SSc; Limited SSc

SUMMARY:
Eosinophils are involved in tissue remodeling and fibrosis in many inflammatory diseases. Systemic sclerosis (SSc) is an autoimmune disease with fibrotic skin and lung complications. The profibrosing properties and data from the SSc literature suggest a possible role of the eosinophils in the process of fibrogenesis of SSc.

DETAILED DESCRIPTION:
it will assess the activation state of blood eosinophils in SSc patients compared to healthy controls (ECP production in vitro, surface activation markers, whole transcriptome array, ..).

it will also study skin eosinophils and their recruitment (extracellular eosinophil granules, eotaxins production in skin, ..)

ELIGIBILITY:
Inclusion Criteria:

* For SSc patients:
* Meeting the 2013 ACR-EULAR criteria for diffuse SSc (n = 20) and limited SSc (n = 20)
* Having signed the informed consent
* Eosinophils ≥ 0.1 G / L on the last blood test (<3 months)

For healthy subjects:

* Without chronic pathology requiring long-term treatment
* Eosinophils between 0.1 and 0.4 G / L on recent blood test (<3 months)

Exclusion Criteria for patients and controls:

* Patient with an infection, state of emergency or progressive neoplastic pathology
* Pregnant or lactating women
* History of atopy (allergic asthma, atopic eczema, allergic rhinitis, allergic conjunctivitis)
* Allergy to local anesthetics (for scleroderma patients only)
* Taking into account a minimum weight of 50 kg and in the absence of cardiorespiratory effects of scleroderma, only patients with at least 10 g of hemoglobin will be included

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The active line of the Internal Medicine department (> 400 sclerodermic patients) guarantees the recruitment of 20 diffuse forms and 20 limited forms
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2018-10-03 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2022-04-05 (Actual)

PRIMARY OUTCOMES:
Comparison of ECP concentrations in supernatants of eosinophils culture | Baseline: one session
  Eosinophils will be sorted, stimulated in vitro for 2 hours and ECP concentration will be assessed in supernatants

SECONDARY OUTCOMES:
Comparison of median fluorescence intensities of several surface markers on blood eosinophils, or comparison of percentages of positive cells among all eosinophils for a given marker (flow cytometry) | Baseline: one session
  MFI/% of CD69, HLA class II, CD9, CD11c, CD44, CCR3, CRTH2, IL-5R on blood eosinophils
Gene expression profiles will be compared between SSc patients and healthy controls (whole transcriptome assay) | Baseline: one session
  Whole genome, transcriptomic approach (differentially expressed genes will be identified using a fold change cutoff)
In skin biopsies: density of eosinophils, extracellular ECP and MBP deposits (absent in healthy skin), and density of eotaxin-1-producing cells will be assessed in damaged skin and apparently healthy skin of SSc patients | Baseline: one session

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Lefevre, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Claude Huriez, CHU, Lille, France